CLINICAL TRIAL: NCT02241343
Title: Venous Occlusion and Limb Swelling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ICREC 13 6 5
Record Dates: First submitted 2014-08-05; First posted 2014-09-16 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Venous Occlusion
Keywords: Venous occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial cohort (Other): Measurements taken before and after venous occlusion applied
  Interventions: Device: Venous occlusion (leg tourniquet, made in-house)

INTERVENTIONS:
Device: Venous occlusion (leg tourniquet, made in-house) — Leg occlusion applied via a blood pressure cuff. Venous occlusion checked using duplex ultrasound

SUMMARY:
Problems affecting the veins in the legs can cause discomfort and swelling. We want to see how artificially and reversibly blocking the leg veins affects swelling in the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, able to consent

Exclusion Criteria:

* History of cardiovascular/renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Trial Cohort: All participants
Period: Overall Study
Arm/Group | Trial Cohort
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trial Cohort
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Leg Swelling
Description: Perometer measured leg volume from footplate to middle of knee joint (in standing position; ml)
Time Frame: 30 minutes
Population: Adverse event precluded data collection
Arm/Group | Trial Cohort
Number analyzed (Participants) | 0

2. Secondary Outcome: Venous Diameter
Description: Great saphenous vein diameter at the knee, taken with duplex ultrasound (cm)
Time Frame: 30 minutes
Population: Zero analysed due to adverse event during protocol
Arm/Group | Trial Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Trial Cohort
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trial Cohort (N=1)
Faint (Investigations) | 1 (1) — Subject fainted shortly after venous tourniquet applied. Reduction in venous return thought to adversely affect perfusion. Fully recovered after release of tourniquet. No injuries sustained

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes